CLINICAL TRIAL: NCT06303232
Title: Combined Effects of Manual Lymphatic Drainage and Therapeutic Ultrasound on Breast Engorgement, Pain and Self Efficacy in Postpartum Women
Brief Title: Effects of Manual Lymphatic Drainage and Therapeutic Ultrasound on Breast Engorgement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0578
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Postpartum Complication
Keywords: Breast engorgement; manual lymphatic drainage; therapeutic ultrasound; pain; self-efficacy; post - partum women.
MeSH Terms: conditions — Pain | interventions — Manual Lymphatic Drainage; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MANUAL LYMPHATIC DRAINAGE (Experimental)
  Interventions: Other: MANUAL LYMPHATIC DRAINAGE
- THERAPEUTIC ULTRASOUND (Active Comparator)
  Interventions: Other: THERAPEUTIC ULTRASOUND

INTERVENTIONS:
Other: MANUAL LYMPHATIC DRAINAGE — MLD was performed after the moist heating of 10 minutes in supine position with both knees bent. It will start from the abdominal lymph drainage followed by the central lymph drainage.
  Then, by stimulating the bilateral axillary lymph nodes, the flow of the fluid was directed to the axillary lymph node. Each session lasted for approximately 45 minutes, for 7 days
  Arms: MANUAL LYMPHATIC DRAINAGE
Other: THERAPEUTIC ULTRASOUND — The participants of group B will receive a treatment of manual lymphatic drainage and ultrasound after the moist heat of 10 minutes. After MLD of 45 minutes, ultrasound will be performed in small circular pattern from periphery to the center towards the areola with following parameters: Mode: pulsed, Frequency: 1MHz, Intensity: 1W/cm2, Time: 8 minutes. Treatment was given for 7 consecutive days
  Arms: THERAPEUTIC ULTRASOUND

SUMMARY:
To find the combined effects of the manual lymphatic drainage with therapeutic ultrasound on breast engorgement, pain and self-efficacy in post - partum women.

ELIGIBILITY:
Inclusion Criteria:

* Both primiparous or multiparous breastfeeding women
* BMI: ≤30-≥25 (14)
* Immediate puerperium with normal or C - section non-premature childbirth (19)
* Postnatal lactating mother with symptoms of breast engorgement

Exclusion Criteria:

* any breast infection, abscess, mastitis, breast cancer
* torn/bleeding or crack nipples
* any skin condition like dermatitis, psoriasis etc
* non-lactating mothers
* having heart pacemaker

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — POST - PARTUM WOMEN
Enrollment: 42 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale - VAS | 7th day
  VAS is an effective rule is measuring the pain score. It ranges from 0 -10 cm line scale with the following description; 0 cm = no pain
  1 - 3 cm = mild pain 4 - 7 cm = moderate pain 8 - 10 cm = severe pain (20). When assessing the validity of VAS, a good-to-excellent correlation was found (r = 0.941), this scale had excellent test-retest reliability. The intra - class correlation coefficients of the VAS was 0.97
Six Point Engorgement Scale - SPE | 7th day
  Six point engorgement scale was the scale for the determination of the breast engorgement.
  The reliability of tool engorgement was 0.948 (22). The score of this scale ranges from 1 - 6.
  Every score has a following description;
  1. = no changes in breast / soft breast
  2. = slight changes in breast
  3. = firm but no breast tenderness
  4. = firm with starting breast tenderness
  5. = tender and firm
  6. = very tender and very firm
Breastfeeding Self-Efficacy Scale - BSES | 7th day
  It includes the 14 items that measure the confidence of the breastfeeding. The divergent validity of the BSES-SF was proved via a significant negative correlation with scores of the Edinburgh Postnatal Depression Scale (r = - 0.273, P < 0.001). In sum, BSES-SF is a reliable and valid instrument for measuring breastfeeding self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: hina gul gul, phd*, Principal Investigator — Riphah International University
Locations (1):
- Innovative Health Concepts Clinic, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lyons KE, Ryan CA, Dempsey EM, Ross RP, Stanton C. Breast Milk, a Source of Beneficial Microbes and Associated Benefits for Infant Health. Nutrients. 2020 Apr 9;12(4):1039. doi: 10.3390/nu12041039. PMID 32283875
- [Background] Mitchell KB, Johnson HM. Breast conditions in the breastfeeding mother. Breastfeeding: Elsevier; 2022. p. 572-93.
- [Background] Napisah P, Widiasih R, Maryati I, Hermayanti Y, Natasya W. The effectiveness of cabbage leaf compress and the education of lactation management in reducing breast engorgement in postpartum. Open Access Macedonian Journal of Medical Sciences. 2021;9(T6):106-10.
- [Background] Indrani D, Sowmya M. A study to find the prevalence of breast engorgement among lactating Mothers. J Reprod Med Gynecol Obstet. 2019;4:023
- [Background] Aprilina HD, Krislinggardini K, Isnaini N, Suratmi S. The effect of cabbage leaves compress on breast engorgement in postpartum mother. Open Access Macedonian Journal of Medical Sciences. 2021;9(T4):124-8
- [Background] Zutshi K, Aman I, Sachdeva T, Khatoon R. Physiotherapy Approach to Breast Engorgement: A Systematic Review. International Journal of Advanced Research in Gynaecology and Obstetrics. 2023;1(1):34-8.
- [Background] Varghese B, Patwa A. Effectiveness of hospital based teaching programme on knowledge regarding home management for breast engorgement among postnatal mothers. Int J Res Rev. 2020;7:486-93.